CLINICAL TRIAL: NCT02471846
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of GDC-0919 Administered With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of GDC-0919 and Atezolizumab Combination Treatment in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29779; 2015-001741-88 (EudraCT Number)
Record Dates: First submitted 2015-06-04; First posted 2015-06-15 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — atezolizumab; navoximod

ARMS (6):
- Anti-PD-1/PD-L1 Relapsed Cohort I (Experimental): Approximately 20 participants whose most recent anti-cancer therapy consisted of single-agent programmed death-1 (PD-1)/programmed death-ligand 1 (PD-L1) blockade and achieved best response of confirmed complete or partial response, or stable disease will receive GDC-0919, at the MTD or maximum administered dose (MAD) determined during the dose-escalation stage, in combination with atezolizumab. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919
- Anti-PD-1/PD-L1 Relapsed Cohort II (Experimental): Approximately 20 participants whose most recent anti-cancer therapy consisted of single-agent PD-1/PD-L1 blockade and achieved unconfirmed partial response or stable disease will receive GDC-0919, at the MTD or MAD determined during the dose-escalation stage, in combination with atezolizumab. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919
- Biopsy Cohort A (Experimental): Approximately 20 participants with melanoma, HNSCC, gastric, ovarian, Merkel cell, cervical, or endometrial cancer will receive GDC-0919 during Cycle 1, followed by combination treatment with GDC-0919 and atezolizumab from Cycle 2 onwards. Serial biopsies of extrahepatic lesions will be performed. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919
- Biopsy Cohort B (Experimental): Approximately 20 participants with melanoma, HNSCC, gastric, ovarian, Merkel cell, cervical, or endometrial cancer will receive atezolizumab during Cycle 1, followed by combination treatment with GDC-0919 and atezolizumab from Cycle 2 onwards. Serial biopsies of extrahepatic lesions will be performed. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919
- Dose-Escalation Cohort(s) (Experimental): Approximately 6 to 65 participants will be enrolled and treated at escalating doses of GDC-0919 in combination with fixed-dose atezolizumab. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio. Successive groups of at least 3 participants will be evaluated during a 21-day window for DLTs, which will determine the enrollment and dosing for subsequent cohorts in the dose-escalation stage. The MTD or MAD, whichever is reached first, will be considered for the expansion stage.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919
- Expansion Cohorts (Experimental): Approximately 160 participants (40 per diagnosis) with NSCLC, RCC, TNBC, and UBC will receive GDC-0919, at the MTD or MAD determined during the dose-escalation stage, in combination with Atezolizumab. Treatment may continue until unacceptable toxicity or disease progression with an unfavorable risk-benefit ratio.
  Interventions: Drug: Atezolizumab; Drug: GDC-0919

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab at a fixed dose of 1200 milligrams (mg) via intravenous (IV) infusion on Day 1 of each 21-day cycle with the exception of biopsy cohort A, where atezolizumab administration will start on Cycle 2 Day 1.
  Other Names: Tecentriq; MPDL3280A; RO5541267
Drug: GDC-0919 — Participants will receive GDC-0919 by mouth (PO) twice daily (BID), specifically every 12 hours. During the dose-escalation stage, the first cohort will receive GDC-0919 at a starting dose of 50 mg PO BID. Dosing will commence on Day -1 for Cycle 1 and follow subsequent 21-day (Days 1 to 21) dosing cycles. The dose will be modified based upon evaluation of DLTs, with single dose escalations not to exceed 2.5-fold of the previous dose. The proposed dosages for evaluation are 50, 100, 200, 400, 600, and 1000 mg PO BID. During the expansion stage, selected solid tumor types will be treated at the MTD or MAD as determined during the dose-escalation stage.

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of the combination of GDC-0919 and atezolizumab in participants with locally advanced, recurrent, or metastatic incurable solid malignancy that has progressed after available standard therapy or for which standard therapy is ineffective, intolerable, or inappropriate. Participants will be enrolled in two stages, including a dose-escalation stage and an expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 12 weeks
* Adequate hematologic and end organ function
* Negative pregnancy test and willingness to utilize contraception among women of childbearing potential
* Locally advanced, recurrent, or metastatic incurable solid malignancy with measurable disease per RECIST v1.1
* Progression following at least one standard therapy; or standard therapy considered ineffective, intolerable, or inappropriate; or use of an investigational agent recognized as a standard of care
* For the expansion stage, histologically confirmed renal cell cancer (RCC), urothelial bladder cancer (UBC), triple-negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), melanoma, head and neck squamous cell carcinoma (HNSCC), gastric cancer, ovarian cancer, cervical cancer, endometrial cancer, or Merkel cell cancer
* For the expansion stage, evaluable for PD-L1 expression
* Anti PD-1/PD-L1 relapsed cohorts (I and II), participants whose most recent anti-cancer therapy consisted of single-agent PD-1/PD-L1 blockade will be enrolled

Exclusion Criteria:

* Significant cardiovascular or liver disease
* Major surgery within 28 days of study drug
* Any anti-cancer therapy within 3 weeks of study drug
* Malabsorption syndrome or poor upper gastrointestinal integrity
* Primary central nervous system (CNS) malignancy or active metastases within 5 years
* Uncontrolled tumor pain
* Autoimmune disease other than stable hypothyroidism or vitiligo
* Human immunodeficiency virus (HIV), active hepatitis B or C, or tuberculosis
* Signs/symptoms of infection, or use of antibiotics within 2 weeks of study drug
* Live attenuated vaccine within 4 weeks of study drug
* Known history or predisposition to QT interval prolongation
* Prior cancer immunotherapy, specifically indoleamine 2,3-dioxygenase (IDO) or tryptophan 2,3-dioxygenase (TDO) inhibitors, T-cell costimulatory receptor agonist antibodies, or checkpoint inhibitors among certain participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-limiting Toxicities (DLTs) | From Day -1 to 21 of Cycle 1 (each cycle is 21 days)
Percentage of Participants With Adverse Events | From Screening until new anti-cancer therapy or up to 60 days after last dose (up to approximately 3 years)

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of GDC-0919 | From Day -1 to 21 of Cycle 1 (each cycle is 21 days)
Recommended Phase II Dose (RP2D) for GDC-0919 | From Day -1 to 21 of Cycle 1 (each cycle is 21 days)
Number of Treatment Cycles Received With GDC-0919 and Atezolizumab | From Day -1 of Cycle 1 (each cycle is 21 days) until treatment discontinuation (up to approximately 3 years)
Dose Intensity of GDC-0919 and Atezolizumab | From Day -1 of Cycle 1 (each cycle is 21 days) until treatment discontinuation (up to approximately 3 years)
Percentage of Participants With Anti-therapeutic Antibody (ATA) Response to Atezolizumab | Pre-dose from Day 1 of Cycle 1 (each cycle is 21 days) up to 120 days after last dose of atezolizumab (up to approximately 3 years)
Plasma Maximum Concentration (Cmax) of GDC-0919 | Post-dose on Day -1 of Cycle 1 (each cycle is 21 days) and Day 1 of Cycle 2
Plasma Minimum Concentration (Cmin) of GDC-0919 | Pre-dose from Day -1 of Cycle 1 (each cycle is 21 days) through Day 1 of Cycle 8
Area Under the Concentration-time Curve to the Last Measurable Concentration (AUC0-last) of GDC-0919 | Pre-dose and post-dose from Day -1 of Cycle 1 (each cycle is 21 days) through Day 1 of Cycle 8
Time to Maximum Concentration (Tmax) of GDC-0919 | Post-dose on Day -1 of Cycle 1 (each cycle is 21 days) and Day 1 of Cycle 2
Serum Cmax of Atezolizumab | Post-dose from Day 1 of Cycle 1 (each cycle is 21 days) up to 120 days after last dose of atezolizumab (up to approximately 3 years)
Serum Cmin of Atezolizumab | Pre-dose from Day 1 of Cycle 1 up to 120 days after last dose of atezolizumab (up to approximately 3 years)
Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as Determined by the Investigator | From Screening until disease progression, death, new anti-cancer therapy, or premature study withdrawal (up to approximately 3 years)
Duration of Objective Response According to RECIST v1.1 as Determined by the Investigator | From Screening until disease progression, death, new anti-cancer therapy, or premature study withdrawal (up to approximately 3 years)
Percentage of Participants With Objective Response According to Modified RECIST as Determined by the Sponsor | From Screening until disease progression, death, new anti-cancer therapy, or premature study withdrawal (up to approximately 3 years)
Duration of Objective Response According to Modified RECIST as Determined by the Sponsor | From Screening until disease progression, death, new anti-cancer therapy, or premature study withdrawal (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (10):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - The Angeles Clinic and Research Institute, Santa Monica Office, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- France (2):
  - Hopital Nord AP-HM, Marseille
  - Institut Gustave Roussy, Villejuif
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Jung KH, LoRusso P, Burris H, Gordon M, Bang YJ, Hellmann MD, Cervantes A, Ochoa de Olza M, Marabelle A, Hodi FS, Ahn MJ, Emens LA, Barlesi F, Hamid O, Calvo E, McDermott D, Soliman H, Rhee I, Lin R, Pourmohamad T, Suchomel J, Tsuhako A, Morrissey K, Mahrus S, Morley R, Pirzkall A, Davis SL. Phase I Study of the Indoleamine 2,3-Dioxygenase 1 (IDO1) Inhibitor Navoximod (GDC-0919) Administered with PD-L1 Inhibitor (Atezolizumab) in Advanced Solid Tumors. Clin Cancer Res. 2019 Jun 1;25(11):3220-3228. doi: 10.1158/1078-0432.CCR-18-2740. Epub 2019 Feb 15. PMID 30770348